CLINICAL TRIAL: NCT03696589
Title: Feasibility and Acceptability of a Physical Activity Behavior Change Intervention for Improving Self-efficacy, Automaticity, and Physical Activity Levels in People With Parkinson's Disease
Brief Title: Feasibility and Acceptability of a Physical Activity Behavior Change Intervention for Parkinson's Disease
Acronym: Preactive-PD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Teachers College, Columbia University (Other)
Responsible Party: Principal Investigator, Lori Quinn, Associate Professor, Teachers College, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-345
Record Dates: First submitted 2018-09-10; First posted 2018-10-04 (Actual); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-08

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single arm cohort study with pre and post intervention assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Physical Activity Coaching — Based in the self-determination theory, participants will be coached on beneficial exercises, how to utilize supports and overcome barriers to PA engagement. Emphasis of exercise coaching will be on increasing aerobic exercise engagement and will include us of Fitbit devices to facilitate uptake and monitor aerobic exercise. Intervention will be delivered by a physical or occupational therapist, who will work with the participant to develop a plan, set goals and targets, and track changes. Additional resources that will support exercise engagement will be provided. Participants will have the choice to receive their face-to-face session either in person or remotely via secure video-based service.

SUMMARY:
The purpose of this study is to assess the feasibility, in regards to acceptability and implementation, of the Pre-Active PD intervention for increased high intensity goal-directed aerobic exercise engagement in people with early-stage Parkinson's disease (Hoehn and Yahr stage I & II). In addition, the study aims to explore the effect estimates of the Pre-Active PD intervention on self-efficacy, motivation, stage of behavior change, and physical activity levels in people with early stage Parkinson's disease.

DETAILED DESCRIPTION:
The investigators will recruit 14 individuals with early stage Parkinson's disease (Hoehn and Yahr stage I & II). The investigators will conduct a single arm cohort. (pre and post intervention) pilot feasibility study over 4 months with embedded process analyses of Preactive-HD, a physical activity coaching intervention program. Previous studies conducted by the investigators will be utilized to adapt the Engage-HD physical activity coaching program to people with early stage PD. The intervention will include a participant/coach interaction and disease-specific workbook grounded within the framework of self-determination theory. The coaching sessions will be conducted by an occupational therapist and will entail six coaching sessions (either face-to-face or remote video sessions via secure Webex connection via computer or smart phone, or phone call if internet/smart phone is not available to participant). The first session (approximately 45 min) will lay the groundwork for the program, and the remaining sessions will serve to provide directed support in relation to regular physical activity and exercise. Participants will develop physical activity goals and will be supported with individual physical activity progression. Participants will be given Fitbit devices as a motivational tool and to track activity progression.

ELIGIBILITY:
Inclusion Criteria:

1. Neurologist confirmed clinical dx for Parkinson's disease Hoehn & Yahr stage I or II
2. Ambulatory for indoor and outdoor mobility without assistance or assistive device
3. Successful completion of Physical Activity Readiness Questionnaire (PAR-Q) (Thomas et al., 1992), or medical clearance from GP

Exclusion Criteria:

1. Musculoskeletal injury that would prevent participation in an exercise program
2. Other neurological disease or disorder such as stroke
3. Already engaging in aerobic exercise for at least 30 minutes for 5 or more days per week.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Quinn, EdD, PT, Principal Investigator — Teachers College, Columbia University
Locations (1):
- Teachers College, Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Coaching: Individuals received 6 sessions of physical activity coaching, delivered either in person or remotely via telehealth
Period: Overall Study
Arm/Group | Physical Activity Coaching
Started | 13
Completed | 12
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Physical Activity Coaching
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.69 (9.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Hoehn & Yahr [Number; unit: participants] — The Hoehn and Yahr Scale is used to measure how Parkinson's symptoms progress and the level of disability. Stages in this study include 1 (Unilateral involvement only usually with minimal or no functional disability) and 2 (Bilateral or midline involvement without impairment of balance)
  participants
    Stage 1 | 4
    Stage 2 | 9
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: units] — The MoCA is a 30-point cognitive screening instrument (scores range from 0-30, with 30 being normal cognitive functioning). A score of less than or equal to 26 is indicative of cognitive impairment.
  units | 27 (3)
URICA-E2 [Mean (Standard Deviation); unit: units] — The URICA-E2 is a 24-item, 5-point Likert-sale, questionnaire. Each item has a statement that reflects an intention toward exercise, with responses ranging from one "strongly disagree" to five "strongly agree". Subscores are used to calculate a Readiness for Change, with possible scores ranging from -2 to +14. Scores of 8 or lower classified as People in Precontemplation, 8-11 classified as People in Contemplation, 11-14 classified as People in Preparation or Action.
  units | 10.7 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Moderate-Vigorous Physical Activity Using Actigraph at 4 Months
Description: Measured using Actigraph accelerometer, levels of moderate-vigorous physical activity will be measured, as well as number of steps and sedentary behavior.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: percentage of time
Groups:
- Physical Activity Coaching - Pretest: Baseline Pretest
- Physical Activity Coaching - Posttest: 4 month posttest
Arm/Group | Physical Activity Coaching - Pretest | Physical Activity Coaching - Posttest
Number analyzed (Participants) | 13 | 12
percentage of time
  %moderate-vigorous physical activity | 2.27 (1.83) | 3.16 (2.07)
  %time sedentary | 76.96 (6.55) | 75.74 (4.59)

2. Primary Outcome: Change From Baseline in the Behavioural Regulation In Exercise Questionnaire (BREQ-2)
Description: The BREQ-2 is a 19-item questionnaire that measures each of the subscales of the self-determination continuum: external, introjected, identified, and intrinsic regulations, as well as amotivation. Each subscale is represented by 4 questions, except for introjected regulation which has 3. Questions are scored using a 5-point Likert scale; Answers range from 0 (not true for me) to 4 (very true for me). Composite scores were calculated from these subscales. Autonomous motivation was calculated from the intrinsic motivation and identified regulation subscales, with possible scores ranging from 0 (low autonomous motivation) to 4 (high autonomous motivation. Controlled motivation was calculated from the introjected regulation and external regulation subscales, with possible scores ranging from 0 (low controlled motivation) to 4 (high controlled motivation).
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Physical Activity Coaching - Pretest: Baseline pre-test assessment
- Physical Activity Coaching - Posttest: 4 month Post-test assessment
Arm/Group | Physical Activity Coaching - Pretest | Physical Activity Coaching - Posttest
Number analyzed (Participants) | 13 | 12
score on a scale
  Controlled motivation | 1.28 (0.86) | 1.56 (0.74)
  Autonomous motivation | 3.16 (0.68) | 3.23 (0.58)

3. Secondary Outcome: Change From Baseline Timed-up-and-go (TUG) at 4 Months
Description: Participant starts sitting in chair and then rises when prompted to "go" and then walks 3 meters, turns around, and walks back to chair. Time to complete is recorded
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Physical Activity Coaching Pretest: Baseline pretest
- Physical Activity Coaching Posttest: 4 months posttest
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
seconds | 7.34 (2.79) | 7.67 (1.50)

4. Secondary Outcome: Change From Baseline 6 Minute Walk Test at 4 Months
Description: Assesses the distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
meters | 461.42 (79.22) | 442.96 (87.61)

5. Secondary Outcome: Change From Baseline Brunel Lifestyle Inventory at 4 Months
Description: The Brunel lifestyle inventory is a 10-item questionnaire that measures both pre-planned (6 items) and un-planned (3 items) lifestyle PA. Scoring for each item is on a scale of 1-5, and the scores for each subscale are averaged. Scores range from 1 (low level of physical activity) to 5 (high level of physical activity).
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
score on a scale
  Planned physical activity | 3.79 (0.78) | 4.14 (0.77)
  Unplanned physical activity | 2.31 (0.67) | 2.56 (0.77)

6. Secondary Outcome: Change From Baseline Wechsler Adult Intelligence Scale -III (WAIS-III) Digit Span Forward and Backward at 4 Months
Description: This test evaluates the number of digits a person can remember in both a forward and backward recall. WAIS-III subscale measures sequential processing, mental manipulation, attention, concentration, memory span, and short-term auditory memory. Higher numbers would indicate a greater number of digits remembered (better outcome). Minimum value is 0 and there is no maximum.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: digits
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
digits | 10.33 (3.31) | 11.27 (2.83)

7. Secondary Outcome: Change From Baseline Stroop Color-Word Interference at 4 Months
Description: This test evaluates the ability to state the color of a word but not the written word. The cognitive dimension tapped by the Stroop is associated with cognitive flexibility, resistance to interference from outside stimuli, creativity, and psychopathology. The number of correct words in 45 seconds is recorded.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: correct words
Groups:
- Physical Activity Coaching Pretest: Baseline Pre-test
- Physical Activity Coaching Posttest: 4 months post-test
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
correct words | 38.42 (10.31) | 40.50 (10.72)

8. Secondary Outcome: Change From Baseline Canadian Occupational Performance Measure (COPM) at 4 Months
Description: Designed to capture a client's self-perception of performance in everyday living, over time. Participants rate their performance and satisfaction of previously defined goals on a scale of 1-10, with 10 being high performance or satisfaction, and 1 being low performance or satisfaction.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
units on a scale
  Performance | 4.99 (1.89) | 8.08 (0.89)
  Satisfaction | 5.75 (1.09) | 8.33 (1.09)

9. Secondary Outcome: Change From Baseline Exercise Self Efficacy Questionnaire at 4 Months
Description: 18-item test that measures an individual's self-efficacy to participate in exercise when numerous barriers are present, including both social and physical barriers. Total score is calculated by summing the responses to each question. This scale has a range of total scores from 0-90. A higher score indicates higher self-efficacy for exercise.
Time Frame: baseline and 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Coaching Pretest | Physical Activity Coaching Posttest
Number analyzed (Participants) | 13 | 12
score on a scale | 61.92 (16.89) | 67.42 (13.04)

10. Secondary Outcome: Perceived Autonomy Support Healthcare Climate Questionnaire (HCCQ) at 4 Months
Description: The Perceived Autonomy Support Healthcare Climate Questionnaire is from the Health-Care, Self-Determination Theory Questionnaire Packet that was designed to assess constructs encompassed within Self-Determination Theory (SDT) as it applies to health-care behavior. This is a measure of acceptability of the intervention administered only the 4 month assessment. Scores on this 15-item questionnaire are calculated by averaging the individual item scores, which are rated on a 1-7 Likert scale. Scores range from 1-7, with higher average scores (7 max) represent a higher level of perceived autonomy support.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Coaching Posttest
Number analyzed (Participants) | 12
score on a scale | 6.69 (0.46)

11. Secondary Outcome: Semi-Structured Post-intervention Questionnaire
Description: This purpose developed post-intervention questionnaire will evaluate participant's perceptions of the intervention. Informed by the Theoretical Framework of Acceptability, the questionnaire was designed to inductively evaluate the retrospective acceptability of the intervention. Score on Likert scale 1-5, with 5 being most acceptable.
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Physical Activity Coaching Posttest: 4 month posttest
Arm/Group | Physical Activity Coaching Posttest
Number analyzed (Participants) | 12
units on a scale | 4.35 (0.27)

ADVERSE EVENTS:
Time Frame: 4 months per participant
Arm/Group | Physical Activity Coaching
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03696589/Prot_SAP_000.pdf